CLINICAL TRIAL: NCT05156840
Title: Telehealth for Discharge Outcomes in Children: A Feasibility Study
Brief Title: Telehealth for Discharge Outcomes in Children
Acronym: TeleDOC
Status: Withdrawn | Type: Observational
Why Stopped: No interested participants were recruited within a 4 month period.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1845410
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Hospital Discharge; Telehealth
Keywords: telehealth; hospital discharge; pediatric; telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telehealth: Patients/Caregivers who received a telehealth follow-up visit from a pediatric hospitalist following hospital discharge.
  Interventions: Behavioral: Telehealth follow-up
- Usual Care: Patients/Caregivers who did not receive a telehealth follow-up visit from a pediatric hospitalist following hospital discharge.

INTERVENTIONS:
Behavioral: Telehealth follow-up — A telehealth follow-up visit will be conducted via the Epic electronic medical record with a pediatric hospitalist following hospital discharge.
  Groups: Telehealth

SUMMARY:
This study will test the feasibility of a telehealth follow-up visit for patients and their caregivers who were recently discharged from a general pediatric inpatient unit.

DETAILED DESCRIPTION:
Patient transitions from hospital to home have increasingly become recognized as a critical opportunity to promote patient safety and high quality care, both at University of California Davis Medical Center and nationwide. With over 16,000 children discharged from U.S. hospitals each day and a rate of 1 in 5 experiencing adverse events related to this process, it is estimated that hospital-to-home transition-related adverse events affect over 1.1 million children annually. The quality of hospital discharge also affects hospital readmission rates, length of hospital stay, and parental satisfaction.

Discharge transition difficulties stem largely from care coordination failures throughout the hospital-to-home transition. The investigators recently conducted a qualitative study analyzing perspectives from parents and physicians of 20 children readmitted within 30 days of hospital discharge. The study identified a theme of caregivers having difficulty re-connecting to the child's medical team for ongoing care after discharge. When problems arose, caregivers reported challenges in knowing who to contact, when to reach out for help, and how to navigate the health system to prevent readmission.

The advent of telehealth presents a unique opportunity to provide seamless follow-up for families following hospital discharge. Although telehealth has not previously been studied as a means of providing pediatric follow-up care after hospital discharge, similar methods of providing post-discharge hospital follow-up, including nurse- or physician-led phone calls and nurse home visits, were highly regarded by families, but failed to impact readmission rates. Telehealth provides a unique advantage over these alternate interventions by allowing face-to-face interaction via videoconference between the patient, caregiver, and hospital physician, who is already familiar with the patient's disease course and overall trajectory. At the investigators' site, although telehealth is readily available for use in most any clinical setting, it is not commonly used for hospital discharge follow-up. Therefore, this study proposes to test the feasibility of a telehealth follow-up visit for patients and their caregivers who were recently discharged from a general pediatric inpatient unit.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians of patients recently discharged from the University of California Davis Children's Hospital pediatric hospitalist service, who were offered a telehealth follow-up visit following their child's discharge
* Pediatric hospitalists who discharged the above patients and offered a telehealth follow-up visit following discharge

Exclusion Criteria:

• Parents/legal guardians of children discharged from an intensive care or subspecialty service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will conduct surveys and interviews to evaluate the feasibility of a telehealth follow-up visit between parents/guardians and pediatric hospitalists of children discharged from the University of California Davis Children's Hospital's pediatric hospitalist service. Telehealth follow-up visits will be offered to discharging pediatric patients at the discretion of the pediatric hospitalist who is discharging the patient.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility Objective 1: Telehealth visit offered on hospital discharge | Within 7 days of hospital discharge
  This objective will assess what percentage of patients discharged from the pediatric hospital medicine service were offered a telehealth follow-up visit on hospital discharge.
Feasibility Objective 2: Parent agreement to engage in telehealth visit | Within 7 days of hospital discharge
  This objective will assess what percentage of parents who were offered a telehealth visit following hospital discharge agreed to participate.
Feasibility Objective 3: Successful completion of telehealth | Within 14 days of hospital discharge
  This objective will assess what percentage of scheduled telehealth visits were successfully completed, as reported by the involved pediatric hospitalist.
Feasibility Objective 4: Lack of technical issues | Within 14 days of hospital discharge
  This objective will assess what percentage of scheduled telehealth visits had not technical issues, as reported by both the involved pediatric hospitalist and the involved caregiver.
Feasibility Objective 5: Survey response rates | Within 30 days of hospital discharge
  This objective will assess what percentage of surveys administered to both pediatric hospitalists and caregivers were completed.

SECONDARY OUTCOMES:
Hospital Readmission | Within 30 days of hospital discharge
  This secondary outcome will assess 30-day hospital re-admission rates, by parental report.
Hospital Length of Stay | Within 7 days of hospital discharge
  This secondary outcome will assess hospital length of stay. This information will be extracted from the electronic medical record.
3-Item Care Transitions Measure | Within 30 days of hospital discharge
  This secondary outcome will evaluate parent scores on the 3-item Care Transitions Measure, reflecting on their child's recent care transition from hospital to home. The 3-question survey include 4 answer choices from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicated a better outcome.

IPD SHARING:
Plan to Share IPD: No